CLINICAL TRIAL: NCT03658421
Title: Comparison of Dexmedetomidine as Adjuvant to Different Concentrations of Ropivacaine for Femoral Nerve Blockade in Patients Undergoing Total Knee Arthroplasty
Brief Title: Dexmedetomidine as Adjuvant for FNB in TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Feng Xia, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: [2018]45
Record Dates: First submitted 2018-09-01; First posted 2018-09-05 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Nerve Block; Dexmedetomidine
Keywords: femoral nerve blockade; dexmedetomidine; ropivacaine; anesthesia
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- H group (Experimental): H group stands for High concentration group. A single bolous of 20 ml ropivacaine 0.2% in ultrasound-guided femoral nerve block (FNB) before the TKA surgery, followed by continuous femoral nerve block (CFNB) using ropivacaine 0.2% (5 ml/h) for postoperative analgesia which started right after surgery. After surgery, all patients received multimodal analgesia of 200mg celecoxib every 12 hours. All subjects received anothother intravenous patient-controlled analgesia pump (IV-PCA pump), which included 50 mg morphine in 50 ml saline: bolus 2 mg; lock out time, 15 minutes.
  Interventions: Procedure: ultrasound-guided femoral nerve block; Device: intravenous patient-controlled analgesia pump with morphine; Procedure: Continuous femoral nerve block
- L group (Experimental): L group stands for low concentration group. A single bolous of 20 ml ropivacaine 0.1% in ultrasound-guided femoral nerve block (FNB) before the TKA surgery, followed by continuous femoral nerve block (CFNB) using ropivacaine 0.1% (5 ml/h) for postoperative analgesia which started right after surgery. All subjects received anothother intravenous patient-controlled analgesia pump (IV-PCA pump), which included 50 mg morphine in 50 ml saline: bolus 2 mg; lock out time, 15 minutes.
  Interventions: Procedure: ultrasound-guided femoral nerve block; Device: intravenous patient-controlled analgesia pump with morphine; Procedure: Continuous femoral nerve block
- LD group (Experimental): LD group stands for low concentration group with dexmedetomidine. A single bolous of 20 ml ropivacaine 0.1% plus 2 μg/kg dexmedetomidine in ultrasound-guided femoral nerve block (FNB) before the TKA surgery, followed by continuous femoral nerve block (CFNB) using ropivacaine 0.1% (5 ml/h) for postoperative analgesia which started right after surgery. All subjects received anothother intravenous patient-controlled analgesia pump (IV-PCA pump), which included 50 mg morphine in 50 ml saline: bolus 2 mg; lock out time, 15 minutes.
  Interventions: Drug: Dexmedetomidine; Procedure: ultrasound-guided femoral nerve block; Device: intravenous patient-controlled analgesia pump with morphine; Procedure: Continuous femoral nerve block

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine added to lower concentration of ropivacaine for postoperative analgesia in FNB
  Arms: LD group
Procedure: ultrasound-guided femoral nerve block — ultrasound-guided femoral nerve block, a single bolous of 20 ml ropivacaine (concentration 0.2% for H group or 0.1% for L group) before surgery followed by continuous femoral nerve block using an infusion rate of ropivacaine 0.2% 5 ml/h for postoperative analgesia started right after surgery
  Other Names: FNB
Device: intravenous patient-controlled analgesia pump with morphine — All subjects received intravenous patient-controlled analgesia (IV-PCA) pumps to measure additional morphine consumption, which included 50 mg morphine in 50 ml saline: bolus 2 mg; lock out time, 15 minutes.
  Other Names: IV-PCA pump
Procedure: Continuous femoral nerve block — All the continuous femoral nerve block infusion regimes in the pump were connected to CFNB catheter, which contained only ropivacaine with different concentrations (ropivacaine 0.1% for L group and LD group; ropivacaine 0.2% for H group, 5 ml/h).
  Other Names: CFNB

SUMMARY:
The aim of the study was to find out whether addition of dexmedetomidine to lower concentration of ropivacaine preoperatively in femoral nerve block (FNB) would intensify analgesia and preserve quadriceps muscle strength after TKA.

DETAILED DESCRIPTION:
We designed this study to evaluate whether dexmedetomidine added to lower concentration of ropivacaine for FNB can intensify analgesic effect and meanwhile reduce the possibility of lower limb (or quadriceps) weakness. Three groups were compared: 0.2% ropivacaine (H group), 0.1% ropivacaine (L group) and ropivacaine 0.1% added with 2 μg/kg dexmedetomidine (LD group).

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* scheduled for total knee arthroplasty

Exclusion Criteria:

* refusal to participate in this study
* unicompartmental knee arthroplasty
* BMI > 35 kg/m2
* congnitive or phychiatric history
* refusal of general anesthesia
* contraindication to laryngeal mask airway insertion
* contraindication to peripheral nerve block (localized infections, sepsis, coagulopathy, bleeding diathesis or preexisting lower extremity neurological abnormality)
* allergy to the drugs used

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
Change of manual muscle testing (MMT) over 72 hours postoperatively | 0-72 hours postoperatively
  The MMT grading was recorded from 0 to 5 to measure muscle strength at 6, 12, 24, 36, 48 and 72 hours after surgery.
Change of Timed Up and Go test (TUG) over 72 hours postoperatively | 0-72 hours postoperatively
  TUG test was used to assess the patient's mobility that requires both balance and static. It was measured at 24, 48 and 72 hours after surgery.
Change of numeric rating scales (NRS) over 72 hours postoperatively | 0-72 hours postoperatively
  NRS was used to evaluate postoperative pain control. They were measured at 6, 12, 24, 36, 48 and 72 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Xia Feng, MD. Ph.D, Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Department of Anesthesiology, First affiliated hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marhofer D, Kettner SC, Marhofer P, Pils S, Weber M, Zeitlinger M. Dexmedetomidine as an adjuvant to ropivacaine prolongs peripheral nerve block: a volunteer study. Br J Anaesth. 2013 Mar;110(3):438-42. doi: 10.1093/bja/aes400. Epub 2012 Nov 15. PMID 23161360
- [Derived] Yang X, Kang W, Xiong W, Lu D, Zhou Z, Chen X, Zhou X, Feng X. The Effect Of Dexmedetomidine As Adjuvant To Ropivacaine 0.1% For Femoral Nerve Block On Strength Of Quadriceps Muscle In Patients Undergoing Total Knee Arthroplasty: A Double-Blinded Randomized Controlled Trial. J Pain Res. 2019 Dec 17;12:3355-3363. doi: 10.2147/JPR.S217283. eCollection 2019. PMID 31908520